CLINICAL TRIAL: NCT06491758
Title: Effect of Electrical Stimulation of the Auricular Branch of the Vagus Nerve (ABVN) on Cervical Vagus Nerve Action Potentials Phase 2
Brief Title: ABVN Phase 2-Studying the Effect of Stimulation on the Auricular Branch of the Vagal Nerve
Acronym: ABVN2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Thomas V. Nowak, Professor, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006075899- A
Record Dates: First submitted 2024-06-12; First posted 2024-07-09 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Healthy Subjects (Experimental): Subjects who have no gastric symptoms or conditions
  Interventions: Device: ML1101 Stimulus Isolator; Procedure: Vagal Maneuver
- Gastroparesis Subjects (Experimental): Subjects with a confirmed diagnosis of gastroparesis.
  Interventions: Device: ML1101 Stimulus Isolator; Procedure: Vagal Maneuver

INTERVENTIONS:
Device: ML1101 Stimulus Isolator — Electrical stimulation electrodes will be placed on the ear with the intensity of the current being increased by 10 percent every 60 seconds, the subject will grade the intensity of the current on a scale of 0-10. Increasing of the current will occur until the subject reports a comfortable level. Once the target level has been achieved the stimulation will be delivered for 2 minutes.
Procedure: Vagal Maneuver — Subjects will undergo the following procedures to stimulate the vagus nerve.
  * Cough: 6 to 8 forceful coughs
  * Cold stimulus: a washcloth soaked in ice water will be placed on the face for 10 seconds.
  * Carotid massage
  * Gagging: a tongue depressor will be inserted for 10 seconds into the mouth touching the back of the mouth.
  * Valsalva maneuver: subjects will will be asked to bear down as if they were having a bowel movement. They will be asked to blow through a mouthpiece that is hooked to a machine that measures how hard they are blowing.
  * Eating: Subjects will be asked to drink water ( 8oz or 1 cup) or/ and Ensure Original ( 8 oz or 1 cup) that has 220 calories after fasting overnight to see that effect on vagal activity during eating.

SUMMARY:
The purpose of this study is to find out if we can gain access to the vagus nerve which is largely an internal nerve that controls stomach function. We hope to gain access to the internal vagus nerve by electrically stimulating the nerve around the external ear. If we can do this then we hope that this will help our treatment of patients with nausea and vomiting and disordered stomach function

DETAILED DESCRIPTION:
Subjects will undergo transcutaneous stimulation of the auricular branch of the vagus nerve and also undergo blood draw before, after stimulation and later a third draw after a period of no stimulation. Healthy subjects will also undergo vagal maneuver using the Multi Array Electrodes (MEA). Gastroparetic subjects will also undergo vagal maneuver using either the regular EKG electrodes or the MEA electrodes.

Subjects will also complete health history questionnaires.

ELIGIBILITY:
Inclusion Criteria healthy volunteers

* Healthy volunteers with no gastric symptoms or conditions (except due to COVID 19)
* Aged 18-80 years
* Willing to have electrodes placed in the external ear (ABVN arm)
* Willing to perform vagal activity maneuver (Vagal arm)
* Willing to have 1 tablespoon (15 ml) of blood drawn at 3 time points

Inclusion Criteria gastroparesis subjects

* Gastroparesis subjects with a confirmed diagnosis of gastroparesis from a GI physician
* Have a formal diagnosis of gastroparesis or are seeing the GI physician for symptoms related to gastroparesis
* Aged 18-80 years
* Willing to have electrodes placed in the external ear (ABVN arm)
* Willing to perform vagal activity maneuver (Vagal arm)
* Willing to have 1 tablespoon (15 ml) of blood drawn at 3 time points

Exclusion Criteria:

* Unable to provide consent
* Pregnant females
* Prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Amplitude of vagal nerve compound action | 3 hours
  To measure the amplitude of vagal nerve compound action potentials during stimulation of the auricular branch of the vagal nerve and during vagal maneuvers.
Respiratory Changes in heart rate during stimulation | 3 hours
  To measure respiratory changes in heart rate during stimulation of the auricular branch of the vagal nerve and also during the vagal maneuvers phase.
Changes in amplitude of the surface electrogastrogram | 3 hours.
  To measure the changes of surface electrogastogram during stimulation of the auricular branch of the vagal nerve and also during the vagal maneuvers phase.
Changes in gastric hormones | 3 hours.
  To measure the effect of stimulation of the auricular branch of the vagal nerve and/or of vagal maneuvers on gastric hormones.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas V Nowak, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with other researchers for similar purposes as to this study
Supporting Information: CSR, Analytic Code
Time Frame: Three years after study completion
Access Criteria: None as of yet.